CLINICAL TRIAL: NCT07185178
Title: Investigation of the Effect of Video Game-Based Breathing Exercises on Dysfunctional Respiration in Patients With Asthma-COPD Overlap Syndrome (ACOS)
Brief Title: Effect of Video Game-Based Breathing Exercises on Respiratory Dysfunction in ACOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hg_tez
Record Dates: First submitted 2025-08-03; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-06

CONDITIONS: Asthma-COPD Overlap Syndrome; Pulmonary Rehabilitation; Video Games
Keywords: asthma-copd overlap syndrome; pulmonary rehabilitation; dysfunctional breathing; video games
MeSH Terms: conditions — Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: The group receiving video game-based breathing exercises (Experimental): Participants in the study group will undergo the "Breathing Games" exercise program twice a week for 8 weeks, with each session lasting approximately 50 minutes.
  Interventions: Other: Video game-based breathing exercises
- Group 2: Control group (Experimental): Participants in the control group will receive a 30-45 minute patient education session after the assessment.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Video game-based breathing exercises — Twenty individuals will be enrolled in the video game-based breathing exercise program. Participants in the study group will undergo the "Breathing Games" exercise program twice a week for 8 weeks, with each session lasting approximately 50 minutes. This video game-based breathing exercise program includes warm-up, cool-down, and five breathing games designed for the target patients.From the second week onward, posture exercises combined with the breathing games will be added.Thus, the exercise program will consist of a warm-up phase lasting approximately 10 minutes, including breathing control, stretching exercises, and rest; 25-30 minutes of five breathing games combined with posture exercises; followed by a cool-down phase of about 10 minutes with breathing control, stretching exercises, and rest.Additionally, participants will be provided with a home exercise program to be performed twice daily for 30 minutes, three days a week, over 8 weeks.
  Arms: Group 1: The group receiving video game-based breathing exercises
Other: Control group — Participants in the control group will receive a 30-45 minute patient education session after the assessment. The content of the education will include:
  Providing general information about Asthma-COPD Overlap Syndrome (ACOS) Teaching dyspnea-relieving positions Instruction in diaphragmatic breathing techniques Teaching secretion clearance methods (Active Cycle of Breathing Techniques - ACBT) Educating on energy conservation strategies Providing information on correct posture Counseling on lifestyle modifications (e.g., smoking cessation, physical activity recommendations) To maintain and improve physical activity levels, patients will be advised to engage in walking activities for 30 minutes, twice a week After covering these topics, participants will be given brochures containing this information. Additionally, follow-up will be conducted by phone every two weeks. All assessments will be repeated at the end of the 8-week period.
  Arms: Group 2: Control group

SUMMARY:
Asthma and COPD are significant respiratory diseases that can coexist, referred to as Asthma-COPD Overlap Syndrome (ACOS). Patients with ACOS experience more severe clinical outcomes, including rapid decline in lung function, increased symptom burden, and reduced quality of life. Pulmonary rehabilitation-particularly breathing exercises-is a core non-pharmacological intervention recommended for this patient group. In recent years, video game-based applications have emerged as innovative tools that enhance motivation and participation in exercise programs. However, studies investigating the effects of video game-based breathing exercises in ACOS patients are extremely limited. Additionally, although dysfunctional breathing patterns are common in this group, few studies have addressed targeted interventions. The objective of the present study is to evaluate the effects of video game-based breathing exercises on dysfunctional breathing in ACOS patients.

DETAILED DESCRIPTION:
Asthma and chronic obstructive pulmonary disease (COPD) are significant public health problems. Asthma is defined as a chronic respiratory disease characterized by airway hyperresponsiveness causing intermittent and usually reversible airway obstruction, whereas COPD is a chronic respiratory disease characterized by progressive and irreversible airway obstruction, typically occurring in individuals over the age of 40 and associated with tobacco use. These definitions allow asthma and COPD to be recognized as distinct diseases. However, many epidemiological studies indicate that asthma and COPD can coexist, or that one condition may progress into the other, a condition referred to as Asthma-COPD Overlap Syndrome (ACOS). According to global guidelines, individuals who are generally aged 40 years or older, have a history of smoking at least five pack-years or biomass exposure, have a medical history of asthma or allergy, and show a post-bronchodilator FEV₁ increase of typically 12% and 200 mL are considered to have ACOS. Compared to patients with asthma or COPD alone, those with ACOS tend to experience more frequent exacerbations, rapid decline in lung function, and reduced health-related quality of life. These factors contribute to higher mortality rates among ACOS patients. Reports indicate that ACOS patients experience more dyspnea, higher comorbidity indices, more frequent hospitalizations, and higher BODE indices. Functional exercise capacity has also been found to be lower in this group.

A review of the literature suggests pulmonary rehabilitation as a non-pharmacological treatment method for ACOS patients. Breathing exercises, forming the basis of pulmonary rehabilitation, aim to reduce dyspnea and hyperinflation, improve respiratory muscle performance, and optimize thoraco-abdominal movement by regulating respiratory muscle activation and patterns. The most commonly used breathing exercises include deep diaphragmatic and segmental breathing exercises (also known as breathing control), pursed-lip breathing, and thoracic expansion exercises. Pulmonary rehabilitation applied to individuals with ACOS has been reported to improve functional capacity and BODE index, reduce dyspnea and symptom scores, and contribute to improved lung function. Studies investigating the effectiveness of pulmonary rehabilitation have shown significant improvements in six-minute walk distance, BODE index, and quality-of-life questionnaire results. In COPD and ACOS patients, significant improvements have been observed after training in lung function, six-minute walk test distance, peripheral and inspiratory muscle strength, activities of daily living, and quality-of-life scores. Considering the clinical course, further research is necessary to develop personalized pulmonary rehabilitation programs for ACOS patients.

No studies have been found applying video game-based exercise programs specifically for ACOS patients. Initially incorporated only into exercise training programs, these digital applications have recently been integrated into respiratory exercise regimens due to technological advancements and have been established in the literature as comprehensive, effective, and innovative treatment approaches for respiratory diseases. With advantages such as increasing patient motivation, interest, exercise adherence, and active participation while making exercises more enjoyable, video game-based exercise applications are recognized as effective and beneficial methods. Nonetheless, video game-based respiratory exercise applications remain extremely limited. The current research project implements video game-based breathing exercises in ACOS patients for the first time.

Studies indicate that dysfunctional breathing patterns are common in patients with asthma and COPD. Dysfunctional breathing is a respiratory disorder characterized by irregular breathing patterns, occurring either in the absence of concurrent diseases or secondary to cardiopulmonary conditions. Dysfunctional breathing leads to symptoms such as hyperventilation, dyspnea, increased accessory muscle activity, paradoxical breathing, postural disorders, sleep disturbances, fatigue, and difficulty concentrating. Reports demonstrate that pulmonary rehabilitation reduces symptoms of dysfunctional breathing.

In studies on asthma patients, pulmonary rehabilitation has been reported to have a positive effect on dysfunctional breathing and to improve quality of life as well as anxiety and depression levels. In studies on COPD patients, reductions in dyspnea levels and respiratory symptoms, along with increases in physical activity levels, have been observed. A case study reported that a pulmonary rehabilitation program including breathing and posture exercises improved dysfunctional breathing symptoms, increased breath-holding time, reduced pain and depression findings, and enhanced attention and concentration levels. A review of the literature indicates that studies on dysfunctional breathing are quite limited. Furthermore, no studies have been identified examining dysfunctional breathing in ACOS patients. Therefore, investigating the effects of video game-based breathing exercises on dysfunctional breathing in ACOS patients represents an original contribution.

The objective of the present research is to investigate the effects of video game-based breathing exercises on dysfunctional breathing in patients with ACOS.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 and 80 years
* Diagnosed with Asthma-COPD Overlap Syndrome (ACOS)
* Nijmegen Questionnaire score ≥ 23
* No severe asthma
* No severe COPD
* In a stable condition (no acute exacerbation in the last 4 weeks)
* To have the cognitive level suitable to adapt to video games

Exclusion Criteria:

* Contraindicated for pulmonary rehabilitation
* Diagnosed with cancer
* Having severe cardiovascular disease
* History of thoracic surgery
* Presence of acute infectious disease
* Cognitive impairment
* Presence of vertigo, epilepsy, or visual impairment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Capnography | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  It will be used to evaluate whether ventilation is adequate and if the breathing pattern is appropriate. It is a monitoring device that continuously records the concentration of CO₂ in the exhaled gases during respiration graphically (in mmHg), providing information about the patient's respiratory rate per minute and the amount of CO₂ exhaled in each breath. It measures the partial pressure of CO₂ in the exhaled air, referred to as end-tidal CO₂ (ETCO₂), which is a reliable and time-sensitive clinical measurement of respiratory function. ETCO₂ shows good concurrent validity when compared directly with blood measurements. A value of 35 mmHg or below is commonly used as a cutoff point to define hypocapnia.
Hi-Lo Test | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  This is a clinical assessment used to evaluate the breathing pattern, specifically to determine whether thoracic (chest) or abdominal (diaphragm) movement is more dominant. The patient is seated comfortably, and the clinician stands or kneels slightly to the side in front of the patient. The clinician places one hand on the patient's sternum (breastbone) and the other hand on the upper abdomen (just below the rib cage). This allows the clinician to feel the movements of both the chest and abdominal areas during inhalation. The clinician observes and senses which area moves more with each breath, indicating whether the patient primarily uses chest or abdominal muscles for breathing. Five breathing cycles are assessed.
Manual Assessment of Respiratory Movements (MARM) | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  This method is used to evaluate and measure breathing patterns, particularly the distribution of respiratory movements between the upper and lower parts of the rib cage and the abdomen under various conditions. The 4th and 5th fingers of both hands are placed on the lower ribs, and the vertical and horizontal mobility of the fingers is assessed while the patient breathes in and out.
  If there is more vertical and upper rib cage movement, the upper line will be farther from the horizontal and closer to the apex. If there is more lateral and lower rib cage/abdominal movement, the lower line will be farther from the horizontal and closer to the base.
Posture Assessment - Posture Screen Application | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  Posture examination will be performed using the PostureScreen® Mobile application through a photographic method. This application essentially digitizes a valid posture assessment technique, namely the photographic method using a vertical plumb line or lead wire method. This examination is simple, quick, easily repeatable, and does not require in-depth knowledge of posturology.
  For cervical measurements, forward head tilt, cervical lordosis angle, and lateral deviations of the neck will be evaluated. For thoracic measurements, thoracic kyphosis angle, shoulder height difference, thoracic scoliosis, and scapular position will be assessed.
Nijmegen Questionnaire | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  The Nijmegen Questionnaire is a valid and reliable self-report tool used for the diagnosis of dysfunctional breathing syndrome. Dysfunctional breathing is a disorder characterized by irregular or abnormal breathing patterns, often confused with conditions such as asthma or anxiety. The questionnaire was developed to assess the frequency of respiratory-related symptoms and consists of 16 items in total. These items include clinically relevant symptoms such as shortness of breath, chest pain, dizziness, and tingling sensations. Each item is scored on a scale from 0 (never) to 4 (very often), and the total score provides information about the severity of dysfunctional breathing.

SECONDARY OUTCOMES:
FEV₁ assesment | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  Pulmonary function will be assessed using the Cosmed Micro Quark spirometer in accordance with ATS and ERS criteria. Patients will be informed before the test, which will be performed in a seated position after 15 minutes of rest. With a nasal clip applied and mouthpiece in place, patients will be instructed to take a deep inspiration, exhale forcefully and rapidly, and then inhale deeply again. The test will be repeated three times, and the valid result will be accepted.Forced expiratory volume in one second (FEV₁) will be measured and recorded in liters (L).
Breath-Holding Time Test | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  It is a simple test commonly used to assess respiratory functions. The purpose is to measure how long a person can hold their breath after taking a normal breath
30-Second Sit-to-Stand Test | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  The individual will sit on a chair without armrests, approximately 43 cm high from the ground, with their back straight and feet flat on the floor. Their arms will be crossed over the chest. The test will begin from this position. After the "start" command is given, the individual will be asked to stand up fully and then sit back down repeatedly for 30 seconds. The total number of complete stands performed within 30 seconds will be recorded.
6-Minute Walk Test (6MWT) | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  For the test, patients will be asked to walk as fast as possible at their own pace for six minutes along a 30-meter hospital corridor. The 6MWT will be conducted twice on the same day. Before starting the test, patients will be informed that if they experience excessive shortness of breath, they can rest during the test, and this resting time will be included in the total test duration. During the test, the physiotherapist will walk alongside the patient and encourage them every 30 seconds using standard phrases such as "You're doing very well" or "Keep it up, you're doing great." Heart rate will be monitored before and after the test, and dyspnea perception will be assessed using the Modified Borg Scale (MBS). At the end of the test, the distance walked in six minutes will be recorded.
St. George's Respiratory Questionnaire (SGRQ) | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  The SGRQ is a questionnaire developed by P. Jones in 2009 to assess the health-related quality of life of patients diagnosed with chronic obstructive pulmonary disease (COPD). The questionnaire consists of 50 items divided into three main sections: symptoms (8 items), activity (16 items), and impacts of the disease (26 items) (21). It evaluates respiratory symptoms, activities limited by dyspnea, and the overall effect of the disease on daily life. The total score of the questionnaire ranges from 0 to 100, where 0 indicates no impairment in quality of life, and scores closer to 100 indicate progressively worse quality of life. The validity and reliability study of the scale was conducted in Turkey in 2013 by Polatlı et al. In the reliability analysis of the SGRQ, the Cronbach's alpha internal consistency coefficient was calculated as 0.88 for the entire scale.
Fatigue Severity Scale (FSS) | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  The Turkish validity and reliability of the scale were established by Gencay-Can et al. (2012). The scale consists of 9 items that assess the degree of fatigue experienced over the past week. Each item is scored from 0 (strongly disagree) to 7 (strongly agree), and the total score is calculated by summing all item scores. The highest possible total score is 63. A score of 36 or above indicates the presence of significant fatigue.
Pittsburgh Sleep Quality Index (PSQI) | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  The Turkish validity and reliability of the index were established by Ağargün et al. (1996). The scoring involves 18 items grouped into 7 component scores. Each item is rated on a scale from 0 to 3. The sum of the seven component scores gives the total PSQI score, which ranges from 0 to 21. A higher total score indicates poorer sleep quality. A total PSQI score between 0 and 4 indicates good sleep quality, while a score between 5 and 21 indicates poor sleep quality. Additionally, this reflects serious impairment in at least two components or moderate impairment in three components of the PSQI.
Beck Anxiety Inventory (BAI) | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  The scale was developed by Beck et al. (1988) and adapted into Turkish by Ulusoy et al. (1993). It has been determined to have sufficient reliability and validity. The BAI assesses the frequency of anxiety symptoms experienced by the individual. It is a self-report scale consisting of 21 items, each rated from 0 to 3. The questions ask the patient how much the feelings of distress have bothered them over the past week. The total score ranges from 0 to 63. A higher score on the scale indicates greater severity of anxiety experienced by the individual.
Beck Depression Inventory (BDI) | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  The scale was developed by Beck et al. (1978) and its Turkish adaptation was made by Hisli (1988). It has been determined to have sufficient reliability and validity. It is a self-assessment scale applied to both healthy individuals and psychiatric patient groups. The purpose is to identify the risk of depression and to measure the level and severity changes of depressive symptoms. This form contains a total of 21 self-assessment items and uses a four-point Likert-type scale. Each item is scored from 0 to 3, with increasing severity, and the total score is obtained by summing these scores. A higher total score indicates greater severity of depression.
FEV₁/FVC ratio evaluation | All evaluations will be made to the participants in the first session and will be repeated after 8 weeks.
  Pulmonary function will be assessed using the Cosmed Micro Quark spirometer in accordance with ATS and ERS criteria. Patients will be informed before the test, which will be performed in a seated position after 15 minutes of rest. With a nasal clip applied and mouthpiece in place, patients will be instructed to take a deep inspiration, exhale forcefully and rapidly, and then inhale deeply again. The test will be repeated three times, and the valid result will be accepted.The FEV₁/FVC ratio is used to assess the presence and severity of airway obstruction. This ratio represents the ratio of the volume of air exhaled in one second during forced expiration (FEV₁) to the total forced vital capacity (FVC). The FEV₁/FVC ratio is expressed as a percentage (%).
PEF Assessment | All evaluations will be made to the participants in the first session and will be repeated after 8 weeks.
  Pulmonary function will be assessed using the Cosmed Micro Quark spirometer in accordance with ATS and ERS criteria. Patients will be informed before the test, which will be performed in a seated position after 15 minutes of rest. With a nasal clip applied and mouthpiece in place, patients will be instructed to take a deep inspiration, exhale forcefully and rapidly, and then inhale deeply again. The test will be repeated three times, and the valid result will be accepted.PEF (Peak Expiratory Flow) refers to the maximum airflow rate a person can achieve when exhaling as quickly and forcefully as possible. This measurement is used to assess airway patency and the degree of airway obstruction. PEF is measured in liters per second (L/s).
FEF25-75 assessment | All evaluations will be made to the participants in the first session and will be repeated after 8 weeks.
  Pulmonary function will be assessed using the Cosmed Micro Quark spirometer in accordance with ATS and ERS criteria. Patients will be informed before the test, which will be performed in a seated position after 15 minutes of rest. With a nasal clip applied and mouthpiece in place, patients will be instructed to take a deep inspiration, exhale forcefully and rapidly, and then inhale deeply again. The test will be repeated three times, and the valid result will be accepted.The mean forced expiratory flow (FEF25-75) between 25% and 75% of volumes during forced expiration will be evaluated in liters per second (L/s).
FVC assessment | All assessments will be performed on the participants at the first session and repeated after 8 weeks.
  Pulmonary function will be assessed using the Cosmed Micro Quark spirometer in accordance with ATS and ERS criteria. Patients will be informed before the test, which will be performed in a seated position after 15 minutes of rest. With a nasal clip applied and mouthpiece in place, patients will be instructed to take a deep inspiration, exhale forcefully and rapidly, and then inhale deeply again. The test will be repeated three times, and the valid result will be accepted. Forced vital capacity (FVC) will be measured and recorded in liters (L).

CONTACTS AND LOCATIONS:
Overall Officials: HÜSNA GÜZEL, PT,PhD (c), Principal Investigator — Istinye University; NURGÜL DÜRÜSTKAN ELBASI, asst. prof., Study Director — Istinye University; TUGBA ÖNYILMAZ, asst. prof., Study Chair — Kocaeli University; Haşim Boyacı, Prof. Dr, Study Chair — Kocaeli University
Locations (1):
- Kocaeli University Training and Research Hospital, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
For reasons of participant confidentiality and ethical considerations, sharing of individual participant data (IPD) is not planned for this study.